CLINICAL TRIAL: NCT04497987
Title: A Phase 3 Randomized, Double-Blind, Placebo-Controlled Trial to Evaluate the Efficacy and Safety of LY3819253 Alone and in Combination With LY3832479 in Preventing SARS-CoV-2 Infection and COVID-19 in Skilled Nursing and Assisted Living Facility Residents and Staff; a NIAID and Lilly Collaborative Study
Brief Title: A Study of LY3819253 (LY-CoV555) and LY3832479 (LY-CoV016) in Preventing SARS-CoV-2 Infection and COVID-19 in Nursing Home Residents and Staff
Acronym: BLAZE-2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); AbCellera Biologics Inc. (Industry); Shanghai Junshi Bioscience Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 18063; J2X-MC-PYAD (Other: Eli Lilly and Company); CoVPN #3501 (Other: National Institute of Allergy and Infectious Diseases (NIAID))
Record Dates: First submitted 2020-07-31; First posted 2020-08-04 (Actual); Results first posted 2022-02-04 (Actual); Last update posted 2022-02-04 (Actual); Status verified 2022-02

CONDITIONS: COVID-19; SARS-CoV2
Keywords: Prevention
MeSH Terms: conditions — COVID-19 | interventions — bamlanivimab; etesevimab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (9):
- Bamlanivimab (Part 1) (Experimental): Participants received single Intravenous (IV) infusion of 4200 milligrams (mg) bamlanivimab.
  Interventions: Drug: Bamlanivimab
- Placebo (Part 1) (Placebo Comparator): Participants received single IV infusion of Placebo.
  Interventions: Drug: Placebo
- Bamlanivimab (Part 2-Prevention) (Experimental): Enrollment for Part 2 was not initiated because the efficacy of Bamlanivimab 4200 mg observed in Part 1 significantly diminished the feasibility of enrolling Part 2.
  Interventions: Drug: Bamlanivimab
- Bamlanivimab + Etesevimab (Part 2-Prevention) (Experimental): Enrollment for Part 2 was not initiated because the efficacy of Bamlanivimab 4200 mg observed in Part 1 significantly diminished the feasibility of enrolling Part 2.
  Interventions: Drug: Bamlanivimab; Drug: Etesevimab
- Placebo Comparator: Placebo (Part 2-Prevention) (Placebo Comparator): Enrollment for Part 2 was not initiated because the efficacy of Bamlanivimab 4200 mg observed in Part 1 significantly diminished the feasibility of enrolling Part 2.
  Interventions: Drug: Placebo
- Bamlanivimab (Part 2 - Treatment) (Experimental): Enrollment for Part 2 was not initiated because the efficacy of Bamlanivimab 4200 mg observed in Part 1 significantly diminished the feasibility of enrolling Part 2.
  Interventions: Drug: Bamlanivimab
- Bamlanivimab + Etesevimab (Part 2- Treatment) (Experimental): Enrollment for Part 2 was not initiated because the efficacy of Bamlanivimab 4200 mg observed in Part 1 significantly diminished the feasibility of enrolling Part 2.
  Interventions: Drug: Bamlanivimab; Drug: Etesevimab
- Bamlanivimab (Part 3) (Experimental): Part 3 of the study is exploratory, conducted to study exploratory objectives and is not reported in this record.
  [Participants received single IV infusion of 700 mg bamlanivimab.]
  Interventions: Drug: Bamlanivimab
- Bamlanivimab + Etesevimab (Part 3) (Experimental): Part 3 of the study is exploratory, conducted to study exploratory objectives and is not reported in this record.
  [Participants received single IV infusion of 700 mg bamlanivimab given with 1400 mg etesevimab.]
  Interventions: Drug: Bamlanivimab; Drug: Etesevimab

INTERVENTIONS:
Drug: Bamlanivimab — Administered IV.
  Other Names: LY-CoV555; LY3819253
  Arms: Bamlanivimab (Part 1); Bamlanivimab (Part 2 - Treatment); Bamlanivimab (Part 2-Prevention); Bamlanivimab (Part 3); Bamlanivimab + Etesevimab (Part 2- Treatment); Bamlanivimab + Etesevimab (Part 2-Prevention); Bamlanivimab + Etesevimab (Part 3)
Drug: Placebo — Administered IV.
  Arms: Placebo (Part 1); Placebo Comparator: Placebo (Part 2-Prevention)
Drug: Etesevimab — Administered IV.
  Other Names: LY-CoV016; LY3832479
  Arms: Bamlanivimab + Etesevimab (Part 2- Treatment); Bamlanivimab + Etesevimab (Part 2-Prevention); Bamlanivimab + Etesevimab (Part 3)

SUMMARY:
The purpose of this study is to evaluate whether LY3819253 given alone and with LY3832479 prevent severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection and coronavirus disease - 2019 (COVID-19). Facility staff and residents in contracted skilled nursing and assisted living facility networks with a high risk of SARS-CoV-2 exposure will receive LY3819253, LY3819253 and LY3832479, or placebo via an injection into a vein. Samples will be taken from the nose. Blood samples will be drawn. Participation could last up to 25 weeks and may include up to 19 visits.

ELIGIBILITY:
Inclusion Criteria:

* Part 1 and Part 2: Resident or facility staff in a skilled nursing or assisted living facility with at least one confirmed case of SARS-CoV-2 detection less than or equal to (≤)7 days prior to randomization
* Are men or non-pregnant women who agree to contraceptive requirements
* Agree to the collection of nasal, mid-turbinate, oropharyngeal, and nasopharyngeal swabs, and venous blood as specified in the schedule of activities
* Have venous access sufficient to allow intravenous infusions and blood sampling
* The participant or legally authorized representative give signed informed consent
* Part 3 only: Resident or staff in a skilled nursing or assisted living facility who satisfy at least one of the following at the time of screening

  * Are greater than or equal to (≥) 65 years of age
  * Have a body mass index (BMI) ≥ 35
  * Have chronic kidney disease
  * Have type 1 or type 2 diabetes
  * Have immunosuppressive disease
  * Are currently receiving immunosuppressive treatment, or
  * Are ≥ 55 years of age AND have

    * cardiovascular disease, OR
    * hypertension, OR
    * chronic obstructive pulmonary disease or other chronic respiratory disease
* Positive SARS-CoV-2 test and infusion within 10 days of symptom onset, OR positive SARS-CoV-2 test and infusion within 10 days of testing if asymptomatic

Exclusion Criteria:

* Parts 1 and 2:

  * Recovered from confirmed COVID-19 disease or asymptomatic infection
  * Prior history of a positive SARS-CoV-2 serology test
  * History of convalescent COVID-19 plasma treatment
  * Participation in a previous SARS-CoV-2 vaccine trial or received an approved SARS-CoV-2 vaccine
  * Previous receipt of SAR-CoV-2-specific monoclonal antibodies
* Have any serious concomitant systemic disease, condition or disorder that, in the opinion of the investigator, should preclude participation in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1180 (Actual)
Dates: Start 2020-08-02 (Actual); Primary Completion 2021-01-16 (Actual); Study Completion 2021-05-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (27):
- United States (27):
  - Unv of AL Sch of Med Div of Infectious Diseases, Birmingham, Alabama
  - Care Access Research, Phoenix, Arizona
  - Allergy and Asthma Clin of NW Ark, Bentonville, Arkansas
  - Care Access Research LLC, Huntington Beach, California
  - Alta Bates SMC, Oakland, California
  - University of Colorado-Anschultz Medical Campus, Aurora, Colorado
  - NIAID, Miami, Florida
  - NIAID, Decatur, Georgia
  - Belmont Village Lincoln Park, Lincoln Park, Illinois
  - Family Medicine, Indianapolis, Indiana
  - University of Louisville, Louisville, Kentucky
  - Care Access Rch Lake Charles, Lake Charles, Louisiana
  - Tulane University School of Medicine, New Orleans, Louisiana
  - NIAID - National Institute of Allergy & Infectious Diseases, Bethesda, Maryland
  - Care Access, Boston, Massachusetts
  - St. Paul IDA-CARe, Saint Paul, Minnesota
  - Care Access, Jackson, Mississippi
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Children's Hospital & Medical Center, Omaha, Nebraska
  - Care Access Research - Bronx, The Bronx, New York
  - NIAD, Chapel Hill, North Carolina
  - Valley Medical Primary Care, Centerville, Ohio
  - Univ of Cin College of Med, Cincinnati, Ohio
  - OSU Med Intl Med Houston Ctr, Tulsa, Oklahoma
  - Donahoe Manor, Bedford, Pennsylvania
  - Belmont Village, West Univ, Houston, Texas
  - Burke Internal Medicine and Research, Burke, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- [Derived] Hirsch C, Park YS, Piechotta V, Chai KL, Estcourt LJ, Monsef I, Salomon S, Wood EM, So-Osman C, McQuilten Z, Spinner CD, Malin JJ, Stegemann M, Skoetz N, Kreuzberger N. SARS-CoV-2-neutralising monoclonal antibodies to prevent COVID-19. Cochrane Database Syst Rev. 2022 Jun 17;6(6):CD014945. doi: 10.1002/14651858.CD014945.pub2. PMID 35713300
- [Derived] Kreuzberger N, Hirsch C, Chai KL, Tomlinson E, Khosravi Z, Popp M, Neidhardt M, Piechotta V, Salomon S, Valk SJ, Monsef I, Schmaderer C, Wood EM, So-Osman C, Roberts DJ, McQuilten Z, Estcourt LJ, Skoetz N. SARS-CoV-2-neutralising monoclonal antibodies for treatment of COVID-19. Cochrane Database Syst Rev. 2021 Sep 2;9(9):CD013825. doi: 10.1002/14651858.CD013825.pub2. PMID 34473343
- [Derived] Nathan R, Shawa I, De La Torre I, Pustizzi JM, Haustrup N, Patel DR, Huhn G. A Narrative Review of the Clinical Practicalities of Bamlanivimab and Etesevimab Antibody Therapies for SARS-CoV-2. Infect Dis Ther. 2021 Dec;10(4):1933-1947. doi: 10.1007/s40121-021-00515-6. Epub 2021 Aug 10. PMID 34374951
- [Derived] Cohen MS, Nirula A, Mulligan MJ, Novak RM, Marovich M, Yen C, Stemer A, Mayer SM, Wohl D, Brengle B, Montague BT, Frank I, McCulloh RJ, Fichtenbaum CJ, Lipson B, Gabra N, Ramirez JA, Thai C, Chege W, Gomez Lorenzo MM, Sista N, Farrior J, Clement ME, Brown ER, Custer KL, Van Naarden J, Adams AC, Schade AE, Dabora MC, Knorr J, Price KL, Sabo J, Tuttle JL, Klekotka P, Shen L, Skovronsky DM; BLAZE-2 Investigators. Effect of Bamlanivimab vs Placebo on Incidence of COVID-19 Among Residents and Staff of Skilled Nursing and Assisted Living Facilities: A Randomized Clinical Trial. JAMA. 2021 Jul 6;326(1):46-55. doi: 10.1001/jama.2021.8828. PMID 34081073
- See also: A Study of LY3819253 (LY-CoV555) to Prevent SARS-CoV-2 Infection and COVID-19 in Nursing Home Residents and Staff (BLAZE-2) — https://trials.lillytrialguide.com/en-US/trial/6hAC2UjP12uxz1fFWVGSKC

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This trial was planned as a 3-part study. Part 1 was to evaluate the efficacy and safety of bamlanivimab (BAM) in preventing severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection and coronavirus disease 2019 (COVID-19), compared with Placebo (PBO). Part 2 was to demonstrate superior efficacy of BAM and BAM + ETE over PBO in the prevention of COVID-19. Part 3 was exploratory cohort.
Pre-assignment Details: Enrollment for Part 2 was not initiated because the efficacy of BAM 4200 mg observed in Part 1 significantly diminished the feasibility of enrolling Part 2.
Groups:
- Placebo: Participants received single IV infusion of Placebo.
- 4200 mg Bamlanivimab: Participants received single IV infusion of 4200 milligrams (mg) bamlanivimab.
Period: Overall Study
Arm/Group | Placebo | 4200 mg Bamlanivimab
Started | 592 | 588
Received at Least One Dose of Study Drug | 587 | 588
Prevention Population | 485 | 487
Treatment Population | 68 | 66
Serology Positive | 36 | 35
Completed | 493 | 521
Not Completed | 99 | 67
Not completed — Adverse Event | 1 | 0
Not completed — Death | 21 | 13
Not completed — Lost to Follow-up | 19 | 17
Not completed — Other - as reported by the investigator | 22 | 16
Not completed — Physician Decision | 1 | 0
Not completed — Withdrawal by Subject | 35 | 21

BASELINE CHARACTERISTICS:
Population: All randomized participants who received at least one dose of study drug.
Groups:
- 4200 mg Bamlanivimab: Participants received single IV infusion of 4200 mg bamlanivimab.
- Total: Total of all reporting groups
Arm/Group | Placebo | 4200 mg Bamlanivimab | Total
Number analyzed (Participants) | 587 | 588 | 1175
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.2 (20.3) | 53.4 (20.7) | 52.8 (20.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 443 | 434 | 877
  Male | 144 | 154 | 298
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 36 | 26 | 62
  Not Hispanic or Latino | 551 | 561 | 1112
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 4 | 5
  Asian | 8 | 6 | 14
  Native Hawaiian or Other Pacific Islander | 3 | 2 | 5
  Black or African American | 52 | 48 | 100
  White | 515 | 519 | 1034
  More than one race | 3 | 5 | 8
  Unknown or Not Reported | 5 | 4 | 9
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 587 | 588 | 1175

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With COVID-19
Description: The endpoint for the primary analysis is defined as the first occurrence of coronavirus disease - 2019 (COVID-19), defined as the detection of severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) by reverse transcription - polymerase chain reaction (RT-PCR) AND mild or worse disease severity within 21 days of detection, by Day 57 (8 weeks after randomization). The participant needed to test positive on or prior to week 8, and they needed to develop their symptoms on or after their positive test date, but no later than 21 days after their positive swab OR Week 8, whichever comes first. Logistic regression model was used which includes occurrence of a primary endpoint event as the response variable, and treatment and stratification factors such as facility as explanatory variables.
Time Frame: Week 8 after randomization
Population: All randomized participants from prevention population.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Groups:
- 4200mg Bamlanivimab: Participants received single IV infusion of 4200mg bamlanivimab.
Arm/Group | Placebo | 4200mg Bamlanivimab
Number analyzed (Participants) | 485 | 487
Percentage of Participants | 15.7 [12.5 to 18.9] | 8.3 [5.8 to 10.7]
Statistical Analysis 1: Comparison: Placebo vs 4200mg Bamlanivimab; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 0.40, 95% CI 2-sided [0.26 to 0.63]

2. Secondary Outcome: Percentage of Participants With Moderate or Worse Severity COVID-19
Description: The endpoint defined as the detection of SARS-CoV-2 by polymerase chain reaction (RT-PCR) AND moderate or worse disease severity within 21 days of detection, by Day 57 (Week 8) were summarized by treatment group. The participant needed to test positive on or prior to week 8, and they needed to develop their symptoms on or after their positive test date, but no later than 21 days after their positive swab OR Week 8, whichever comes first. Logistic regression model was used which includes occurrence of a primary endpoint event as the response variable, and treatment and stratification factors such as facility as explanatory variables.
Time Frame: Week 8 after randomization
Population: All randomized participants from prevention population.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Placebo | 4200mg Bamlanivimab
Number analyzed (Participants) | 485 | 487
Percentage of Participants | 14.7 [11.5 to 17.8] | 8.1 [5.6 to 10.5]
Statistical Analysis 1: Comparison: Placebo vs 4200mg Bamlanivimab; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 0.43, 95% CI 2-sided [0.27 to 0.67]

3. Secondary Outcome: Percentage of Participants With SARS-CoV-2
Description: Percentage of Participants with SARS-CoV-2.
Time Frame: Week 4
Population: All randomized participants from prevention population.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Placebo | 4200mg Bamlanivimab
Number analyzed (Participants) | 485 | 487
Percentage of Participants | 23.1 [19.4 to 26.9] | 17.8 [14.4 to 21.2]
Statistical Analysis 1: Comparison: Placebo vs 4200mg Bamlanivimab; Test type: Superiority; p = 0.021, Regression, Logistic; Odds Ratio (OR) = 0.66, 95% CI 2-sided [0.46 to 0.94]

4. Secondary Outcome: Percentage of Participants Who Are Hospitalized or Have Died Due to COVID-19
Description: Percentage of Participants Who are Hospitalized or Have Died due to COVID-19.
Time Frame: Week 8
Population: All randomized participants from prevention population.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Placebo | 4200mg Bamlanivimab
Number analyzed (Participants) | 485 | 487
Percentage of Participants | 1.4 [0.4 to 2.5] | 0.4 [0 to 1.0]

5. Secondary Outcome: Percentage of Participants Who Experience COVID-19-Related Hospitalization, COVID-19 Related Emergency Room Visit, or Death
Description: Percentage of Participants who Experience COVID-19-Related Hospitalization, COVID-19 Related Emergency Room Visit, or Death.
Time Frame: Week 8
Population: All randomized participants from prevention population.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Placebo | 4200mg Bamlanivimab
Number analyzed (Participants) | 485 | 487
Percentage of Participants | 1.4 [0.4 to 2.5] | 0.6 [0 to 1.3]

6. Secondary Outcome: Percentage of Participants Who Die Due to COVID-19
Description: Percentage of Participants Who Die Due to COVID-19.
Time Frame: Week 8
Population: All randomized participants from prevention population.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Placebo | 4200mg Bamlanivimab
Number analyzed (Participants) | 485 | 487
Percentage of Participants | 0.8 [0 to 1.6] | 0 [0 to 0]

7. Secondary Outcome: Pharmacokinetics (PK): Mean Concentration of Bamlanivimab Administered Alone
Description: Pharmacokinetics (PK): Mean Concentration of bamlanivimab Administered Alone.
Time Frame: Day 29, 57, 85, 141 and 169
Population: All randomized participants who received at least one dose of bamlanivimab and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram per milliliter (µg/mL)
Arm/Group | 4200mg Bamlanivimab
Number analyzed (Participants) | 557
microgram per milliliter (µg/mL)
  Day 29 | 162 (44.4)
  Day 57: number analyzed (Participants) | 536
  Day 57 | 61.8 (59.9)
  Day 85: number analyzed (Participants) | 369
  Day 85 | 28.4 (61.6)
  Day 141: number analyzed (Participants) | 137
  Day 141 | 17.5 (46.2)
  Day 169: number analyzed (Participants) | 49
  Day 169 | 15.1 (42.3)

ADVERSE EVENTS:
Time Frame: Baseline, up to 9 Months
Description: All randomized participants who received at least one dose of study drug. Gender specific events only occurring in male or female participants have had the number of participants At Risk adjusted accordingly.
Arm/Group | Placebo | 4200mg Bamlanivimab
All-Cause Mortality (participants affected / at risk) | 21/587 | 13/588
Serious Adverse Events (participants affected / at risk) | 30/587 | 39/588
Other Adverse Events (participants affected / at risk) | 147/587 | 145/588
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Placebo (N=587) | 4200mg Bamlanivimab (N=588)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 3 (3)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 2 (3) | 2 (2)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1) | 1 (1)
Cardiomyopathy (Cardiac disorders) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 1 (1) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1)
Thyrotoxic crisis (Endocrine disorders) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mouth haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophageal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Death (General disorders) | 1 (1) | 1 (1)
Gait disturbance (General disorders) | 0 (0) | 1 (1)
Sudden death (General disorders) | 0 (0) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic cirrhosis (Hepatobiliary disorders) | 0 (0) | 0 (0)
Acquired immunodeficiency syndrome (Infections and infestations) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 0 (0)
Escherichia bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Escherichia urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Groin abscess (Infections and infestations) | 0 (0) | 1 (1)
Osteomyelitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 2 (2)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 3 (3) | 3 (3)
Septic shock (Infections and infestations) | 1 (1) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 5 (6)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Injury corneal (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0)
Multiple injuries (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Open globe injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 1 (1)
Dementia (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Metabolic encephalopathy (Nervous system disorders) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 2 (2)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 2 (2)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1/443 (1) | 0/434 (0)
Depression suicidal (Psychiatric disorders) | 0 (0) | 1 (1)
Mental status changes (Psychiatric disorders) | 0 (0) | 1 (2)
Post-traumatic stress disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 1 (1)
End stage renal disease (Renal and urinary disorders) | 1 (1) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal artery stenosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0)
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0)
Hypovolaemic shock (Vascular disorders) | 1 (1) | 0 (0)
Lymphoedema (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Placebo (N=587) | 4200mg Bamlanivimab (N=588)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1)
Atrial thrombosis (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 1 (1)
Cardiomegaly (Cardiac disorders) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 3 (3)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 2 (3)
Eustachian tube dysfunction (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Excessive cerumen production (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 5 (5)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 0 (0)
Hyperparathyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Eye discharge (Eye disorders) | 0 (0) | 1 (1)
Eye pruritus (Eye disorders) | 1 (1) | 0 (0)
Retinal detachment (Eye disorders) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abdominal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1)
Anal incontinence (Gastrointestinal disorders) | 0 (0) | 0 (0)
Aphthous ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 3 (3) | 3 (3)
Dental caries (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (2)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 2 (3)
Faecaloma (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric disorder (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 3 (3)
Glossodynia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oral pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Asthenia (General disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1)
Face oedema (General disorders) | 1 (1) | 0 (0)
Feeling hot (General disorders) | 0 (0) | 0 (0)
Infusion site haemorrhage (General disorders) | 0 (0) | 1 (1)
Injection site extravasation (General disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1) | 1 (1)
Oedema (General disorders) | 1 (1) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 1 (1)
Puncture site haematoma (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Swelling face (General disorders) | 0 (0) | 1 (1)
Hepatic cirrhosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1) | 0 (0)
Food allergy (Immune system disorders) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Serum sickness (Immune system disorders) | 1 (1) | 0 (0)
Abscess (Infections and infestations) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 3 (3) | 1 (1)
Candida infection (Infections and infestations) | 2 (2) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 1 (1)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 2 (2)
Conjunctivitis (Infections and infestations) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0)
Ear infection (Infections and infestations) | 2 (2) | 2 (2)
Endocarditis (Infections and infestations) | 0 (0) | 1 (1)
Eye infection (Infections and infestations) | 1 (1) | 0 (0)
Fungal infection (Infections and infestations) | 1 (1) | 0 (0)
Gastrointestinal bacterial infection (Infections and infestations) | 0 (0) | 1 (1)
Kidney infection (Infections and infestations) | 1 (1) | 0 (0)
Labyrinthitis (Infections and infestations) | 0 (0) | 1 (1)
Localised infection (Infections and infestations) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1) | 2 (2)
Oral candidiasis (Infections and infestations) | 0 (0) | 1 (1)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0)
Osteomyelitis (Infections and infestations) | 0 (0) | 1 (1)
Pharyngitis streptococcal (Infections and infestations) | 2 (2) | 0 (0)
Pilonidal cyst (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 7 (7) | 2 (2)
Rhinitis (Infections and infestations) | 1 (1) | 1 (1)
Sinusitis (Infections and infestations) | 8 (8) | 2 (2)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 1 (1)
Tooth abscess (Infections and infestations) | 1 (1) | 3 (3)
Tooth infection (Infections and infestations) | 0 (0) | 3 (4)
Urinary tract infection (Infections and infestations) | 20 (22) | 11 (13)
Vaginal infection (Infections and infestations) | 0/443 (0) | 1/434 (1)
Viral infection (Infections and infestations) | 0 (0) | 1 (1)
Animal bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Animal scratch (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 2 (2) | 3 (3)
Fall (Injury, poisoning and procedural complications) | 9 (12) | 6 (6)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Muscle strain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1) | 2 (3)
Soft tissue injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tibia fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Tooth fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vaccination complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Amylase increased (Investigations) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Blood albumin decreased (Investigations) | 0 (0) | 2 (2)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (1) | 1 (1)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0)
Blood glucose increased (Investigations) | 2 (2) | 1 (1)
Blood potassium decreased (Investigations) | 0 (0) | 1 (2)
Blood pressure increased (Investigations) | 1 (1) | 3 (3)
Blood sodium decreased (Investigations) | 1 (1) | 0 (0)
Blood urea increased (Investigations) | 1 (1) | 1 (1)
Brain natriuretic peptide increased (Investigations) | 0 (0) | 1 (1)
Breath sounds abnormal (Investigations) | 0 (0) | 0 (0)
C-reactive protein increased (Investigations) | 1 (1) | 0 (0)
Capillary nail refill test abnormal (Investigations) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 2 (2) | 1 (1)
Haemoglobin increased (Investigations) | 1 (1) | 0 (0)
Hepatic enzyme increased (Investigations) | 0 (0) | 1 (1)
International normalised ratio increased (Investigations) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (1)
Neutrophil count increased (Investigations) | 1 (1) | 0 (0)
Procalcitonin increased (Investigations) | 0 (0) | 0 (0)
Smear cervix abnormal (Investigations) | 0/443 (0) | 1/434 (1)
Troponin increased (Investigations) | 0 (0) | 1 (1)
White blood cell count decreased (Investigations) | 0 (0) | 1 (1)
White blood cell count increased (Investigations) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 3 (4) | 1 (1)
Dyslipidaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Glucose tolerance impaired (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Gout (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperproteinaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Metabolic acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Vitamin b complex deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Vitamin d deficiency (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (4) | 7 (8)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (6) | 5 (5)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Coccydynia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Inguinal mass (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3) | 4 (4)
Sjogren's syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Trochlear dysplasia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/443 (1) | 0/434 (0)
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/144 (1) | 0/154 (0)
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0)
Bell's palsy (Nervous system disorders) | 0 (0) | 1 (1)
Carpal tunnel syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Cubital tunnel syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 6 (6) | 5 (6)
Dizziness postural (Nervous system disorders) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 2 (2)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 2 (2)
Metabolic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 3 (3) | 1 (1)
Tremor (Nervous system disorders) | 0 (0) | 1 (1)
Anorgasmia (Psychiatric disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 2 (2)
Anxiety disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1)
Delusion (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 3 (3)
Generalised anxiety disorder (Psychiatric disorders) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 2 (2) | 1 (1)
Mental status changes (Psychiatric disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1)
Bladder spasm (Renal and urinary disorders) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 2 (2) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 3 (3) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal impairment (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1) | 0 (0)
Breast mass (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 0/443 (0) | 1/434 (1)
Ovarian cyst ruptured (Reproductive system and breast disorders) | 1/443 (1) | 0/434 (0)
Vulvovaginal pruritus (Reproductive system and breast disorders) | 0/443 (0) | 1/434 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Paranasal sinus discomfort (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pharyngeal paraesthesia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Diabetic foot (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 5 (5)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin wrinkling (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0)
Stasis dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 4 (4)
Dental operation (Surgical and medical procedures) | 1 (1) | 0 (0)
Knee arthroplasty (Surgical and medical procedures) | 1 (1) | 0 (0)
Retinopexy (Surgical and medical procedures) | 0 (0) | 1 (1)
Salpingo-oophorectomy unilateral (Surgical and medical procedures) | 1/443 (1) | 0/434 (0)
Sinus operation (Surgical and medical procedures) | 0 (0) | 1 (1)
Spinal laminectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Tooth extraction (Surgical and medical procedures) | 0 (0) | 1 (1)
Aortic arteriosclerosis (Vascular disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Flushing (Vascular disorders) | 2 (2) | 2 (2)
Haematoma (Vascular disorders) | 1 (1) | 1 (1)
Hypertension (Vascular disorders) | 11 (11) | 8 (8)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Lymphoedema (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2021-01-22): https://cdn.clinicaltrials.gov/large-docs/87/NCT04497987/Prot_000.pdf
  • Statistical Analysis Plan (2020-12-07): https://cdn.clinicaltrials.gov/large-docs/87/NCT04497987/SAP_001.pdf